CLINICAL TRIAL: NCT07349771
Title: Phase II Double-Blinded Placebo-Controlled Randomized Trial of CSF-1R Inhibitor, Axatilimab for Prevention of Acute and Chronic GVHD After HLA-Matched Related and Unrelated Donor Allogeneic Stem Cell Transplantation (ABRAXAS)
Brief Title: Axatilimab Plus Standard of Care Therapy for the Prevention of Graft Versus Host Disease Following Allogeneic Hematopoietic Stem Cell Transplantation in Patients With Hematologic Cancer, ABRAXAS Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: MC230810; NCI-2025-09723 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-009803 (Other: Mayo Clinic Institutional Review Board); MC230810 (Other: Mayo Clinic)
Record Dates: First submitted 2026-01-15; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm
MeSH Terms: interventions — Stem Cell Transplantation; axatilimab; Specimen Handling; Cyclophosphamide; Magnetic Resonance Spectroscopy; Mycophenolic Acid; Tacrolimus; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Intervention Model Description: Safety run-in followed by randomized phase II study design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Stage 1 safety run-in (SOC GVHD prophylaxis, axatilimab) (Experimental): Patients undergo SOC allogeneic HCT on day 0 and receive SOC GVHD prophylaxis consisting of cyclophosphamide IV over 1-2 hours on days +3 and +4, tacrolimus starting on day +5 and tapered through day +90 to +100, and mycophenolate mofetil IV or PO TID on days +5 to +35 in the absence of disease progression or unacceptable toxicity. Starting on day +35, patients also receive axatilimab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 14 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo x-ray or CT during screening and blood sample collection and bone marrow aspiration throughout the study. Patients may also undergo CT, MRI, or PET throughout the study and may optionally undergo skin biopsy on study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Axatilimab; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Magnetic Resonance Imaging; Drug: Mycophenolate Mofetil; Procedure: Positron Emission Tomography; Procedure: Skin Biopsy; Drug: Tacrolimus; Procedure: X-Ray Imaging
- Stage 2 arm I (SOC GVHD prophylaxis, axatilimab) (Experimental): Patients undergo SOC allogeneic HCT and receive SOC GVHD prophylaxis plus axatilimab as in stage 1 safety run-in in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo x-ray or CT during screening and blood sample collection and bone marrow aspiration throughout the study. Patients may also undergo CT, MRI, or PET throughout the study and may optionally undergo skin biopsy on study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Axatilimab; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Magnetic Resonance Imaging; Drug: Mycophenolate Mofetil; Procedure: Positron Emission Tomography; Procedure: Skin Biopsy; Drug: Tacrolimus; Procedure: X-Ray Imaging
- Stage 2 arm II (SOC GVHD prophylaxis, placebo) (Placebo Comparator): Patients undergo SOC allogeneic HCT on day 0 and receive SOC GVHD prophylaxis consisting of cyclophosphamide IV over 1-2 hours on days +3 and +4, tacrolimus starting on day +5 and tapered through day +90 to +100, and mycophenolate mofetil IV or PO TID on days +5 to +35 in the absence of disease progression or unacceptable toxicity. Starting on day +35, patients also receive placebo IV over 30 minutes on day 1 of each cycle. Cycles repeat every 14 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo x-ray or CT during screening and blood sample collection and bone marrow aspiration throughout the study. Patients may also undergo CT, MRI, or PET throughout the study and may optionally undergo skin biopsy on study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Magnetic Resonance Imaging; Drug: Mycophenolate Mofetil; Drug: Placebo Administration; Procedure: Positron Emission Tomography; Procedure: Skin Biopsy; Drug: Tacrolimus; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo SOC allogeneic HCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Biological: Axatilimab — Given IV
  Other Names: Anti-M-CSFR Monoclonal Antibody SNDX-6352; Axatilimab-csfr; INCA 034176; INCA 34176; INCA-034176; INCA-34176; INCA034176; INCA34176; Niktimvo; SNDX 6352; SNDX-6352; SNDX6352; UCB6352
  Arms: Stage 1 safety run-in (SOC GVHD prophylaxis, axatilimab); Stage 2 arm I (SOC GVHD prophylaxis, axatilimab)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: CellCept; MMF
Drug: Placebo Administration — Given IV
  Arms: Stage 2 arm II (SOC GVHD prophylaxis, placebo)
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Skin Biopsy — Undergo skin biopsy
  Other Names: Biopsy of Skin
Drug: Tacrolimus — Given tacrolimus
  Other Names: FK 506; FK-506; FK506; Fujimycin; Hecoria; Prograf; Protopic; Tacforius
Procedure: X-Ray Imaging — Undergo x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase II trial studies how well adding axatilimab to standard of care (SOC) therapy works in preventing graft versus host disease (GVHD) following allogeneic hematopoietic stem cell transplantation (HCT) in patients with hematologic cancer. Allogeneic HCT is a procedure in which a person receives blood-forming stem cells (cells from which all blood cells develop) from a genetically similar, but not identical, donor. This is often a sister or brother, but could be an unrelated donor. Sometimes the transplanted cells from a donor can attack the body's normal cells, causing GVHD. Symptoms of GVHD can include yellowing of the skin, mucous membranes, and eyes, skin rash or blisters, dry mouth, or dry eyes. Typically, drugs such as cyclophosphamide, tacrolimus, and mycophenolate mofetil are given after the transplant to help stop GVHD from happening, but these current therapies may negatively affect patient quality of life and newer treatment strategies are needed. Axatilimab is a monoclonal antibody. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens), which may prevent GVHD from developing. Adding axatilimab to SOC therapy may be more effective in preventing GVHD following allogeneic HCT in patients with hematologic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with a history of a hematologic malignancy with a planned myeloablative conditioning (MAC) peripheral blood allogeneic HCT

  * Note: Patients with acute leukemia must be in morphologic complete remission with or without hematologic recovery with ˂ 5% blasts in the bone marrow. Patients with chronic myelomonocytic leukemia (CMML) must have a white blood cell (WBC) count ≤ 10,000 cells/µL and < 5% blasts in the marrow. Patients with ≥ 5% blasts due to a regenerating marrow must contact the protocol chairs for review. Patients with a diagnosis of myelofibrosis require sponsor approval before enrolling
* Patients must be receiving an allograft from a suitable human leukocyte antigen (HLA)-matched sibling or unrelated donor according to transplant center's guidelines (for selection of appropriate donor)
* Karnofsky performance status ≥ 60
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) or total bilirubin ≤ 3.0 x the ULN in the presence of Gilbert's syndrome (obtained ≤ 14 days prior to registration/randomization). If total bilirubin is abnormal (≥ 1.5 x ULN), assess direct bilirubin. NOTE: Patients with Gilbert syndrome and elevated baseline unconjugated (indirect) bilirubin up to 3.0 mg/dL are eligible. Gilbert syndrome should be confirmed by the presence of UGT1A1*28 variant
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 2.5 x ULN (obtained ≤ 14 days prior to registration/randomization)
* Calculated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault formula (obtained ≤ 14 days prior to registration/randomization)
* Negative serum pregnancy test done ≤ 7 days prior to registration/randomization, for persons of childbearing potential only
* Sexually active patients and their partners must use an effective method of contraception associated with a low failure rate prior to study entry and for the duration of study participation and for at least 3 months after the last dose of study drug

  * Note: The following are considered effective contraceptives: oral contraceptive pill; condom plus spermicide; diaphragm plus spermicide; patient or partner surgically sterile; patient or partner more than 12 months postmenopausal; or injectable or implantable agent/device. Male patients should refrain from sperm donation and female patients should refrain from breastfeeding throughout this period
* Provide written informed consent
* Willingness to provide mandatory blood and bone marrow aspirate specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic, and teratogenic effect on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential, and persons able to father a child, who are unwilling to employ adequate contraception
* Any of the following current or prior therapies:

  * Patients receiving a cord blood transplant
  * Patients undergoing a T-cell depleted allogeneic transplantation (using ex vivo CD34 selection, or with serotherapy [antithymocyte globulin or alemtuzumab])
  * Patients undergoing a second allogeneic transplant (after a previous allogeneic transplant)
  * Pre-planned treatment with JAK1/JAK2 inhibitor after transplant
  * Previous exposure to axatilimab
  * Currently participating in any other interventional study
  * Receiving an investigational treatment ≤ 28 days prior to registration/randomization
  * Major surgery ≤ 3 weeks prior to registration/randomization
  * Chemotherapy ≤ 2 weeks prior to registration/randomization unless chemotherapy is part of the pre-transplant conditioning
  * Radiation therapy ≤ 2 weeks prior to registration/randomization unless radiation is part of the pre-transplant conditioning
  * Planned use of donor lymphocyte infusion (DLI) therapy
  * Exception: Use of maintenance regimens as routine clinical care will be permitted but must be declared prior to registration/randomization. The trial does not restrict subsequent treatment after meeting the GVHD-free survival (GFS) endpoint
* Active central nervous system (CNS) involvement by malignant cells
* Leukemia involvement in the CNS ≤ 4 weeks of registration for patients with a history of prior CNS leukemia involvement (i.e., leukemic blasts previously detected in the cerebral spinal fluid)
* History of acute or chronic pancreatitis
* History of myositis
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Patients with active hepatitis B or C

  * Patients with a history of hepatitis B or C are allowed if hepatitis B virus (HBV) deoxyribonucleic acid (DNA) or hepatitis C virus (HCV) RNA are undetectable
* Any known infection with human immunodeficiency virus (HIV), human T-lymphotropic virus-1 (HTLV-1)
* Uncontrolled bacterial, viral, or fungal infections (currently taking medication and with progression or no clinical improvement) at the time of registration/randomization
* Psychiatric illness/social situations that would limit compliance with study requirements
* Diagnosed with another malignancy (other than malignancy for which transplant was performed) ≤ 3 years of registration/randomization, unless previously treated with curative intent and approved by principal investigator (PI) (e.g., but not limited to completely resected basal cell, squamous cell, or ductal carcinoma in situ, or low-risk prostate cancer after curative resection or on watchful waiting). In patients with transformed disease (e.g. aggressive lymphoma evolving from chronic lymphocytic leukemia [CLL], or acute leukemia from myelodysplastic syndrome [MDS]), the original hematological disorder is not considered an exclusion. Cancer treated with curative intent < 3 years previously will not be allowed unless approved by the study chairs
* History of myocardial infarction ≤ 6 months, or New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2033-01-31 (Estimated)

PRIMARY OUTCOMES:
Graft versus host disease (GVHD)-free survival | At 1 year post-transplant
  Rates will be compared between the two arms. A patient will be considered a success for 1-year GVHD-free survival if they are alive without grade 3 or 4 acute or systemic immunosuppression-requiring chronic GVHD at one year post myeloablative allogeneic hematopoietic cell transplantation (HCT).

SECONDARY OUTCOMES:
Cumulative incidence of mild, moderate, and severe chronic GVHD | Up to 1 year post-transplant
  As assessed by National Institutes of Health criteria. Will be estimated in each arm using the competing risk model, with death without chronic GVHD as a competing risk event. Differences between arms will be evaluated using Cox proportional hazard models with competing risk.
Cumulative incidence of systemic corticosteroid requiring chronic GVHD | Up to 1 year post-transplant
  Will be estimated in each arm using the competing risk model, with death without chronic GVHD requiring systemic corticosteroids as a competing risk event. Differences between arms will be evaluated using Cox proportional hazard models with competing risks.
Cumulative incidence of grade II-IV and III-IV acute GVHD | At 100 days and 180 days
  Will be estimated in each arm using the competing risk model, with death without grade II-IV or III-IV acute GVHD as a competing risk events respectively. Differences between arms will be evaluated using Cox proportional hazard models with competing risks.
Cumulative incidence of non-relapse mortality | Up to 1 year post-transplant
  Will be estimated in each arm using the competing risk model, with relapse/progression as a competing risk event. Differences between arms will be evaluated using Cox proportional hazard models with competing risks.
Incidence of primary and secondary graft failure | At 30 days, 60 days, 100 days, 180 days, and 365 days
  Will be estimated in each arm by the number of patients who experience graft failure divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success rate will be calculated. Differences in rates between arms will be evaluated using Fisher's exact test.
Cumulative incidence of relapse/progression of the primary hematologic malignancy | Up to 2 years
  Will be estimated in each arm using the competing risk model, with death without relapse/progression as a competing risk event. Differences between arms will be evaluated using Cox proportional hazard models with competing risks.
Lineage specific chimerism kinetics | At 30 days, 100 days, 180 days, and 365 days
  The percentage of donor versus recipient cells will be evaluated for T cells (CD3+), myeloid cells (CD33+), B cells (CD19+), and NK cells (CD56+) at each time point to assess lineage specific chimerism kinetics. The percentages will be categorized for each cell type as full recipient (≤ 5%), mixed (6-94%), or full donor (≥ 95%). Values will be summarized descriptively (median, range, distribution across categories) and changes across time will be evaluated.
Immune reconstitution | At 30 days, 100 days, 180 days, and 365 days
  Immune profiles (including helper T cells (CD3+ CD4+), cytotoxic T cells (CD3+ CD8+), regulatory T cells (CD3+ CD4+ CD25+ CD127low/-FOXP3+), B cells (CD19+) will be evaluated at each time point to assess immune reconstitution following transplant. Values at each time point will be summarized descriptively (median, range) and changes across time will be evaluated.
Progression-free survival | Up to 2 years post-transplant
  Defined as the time from transplant to the earliest date of documentation of relapse/progression or death due to any cause.
Overall survival | Up to 2 years post-transplant
  Defined as the time from transplant to death due to any cause.
Incidence of adverse events | Up to 2 years post-transplant
  Assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed for each arm to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh Chhabra, MBBS, MS, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials